CLINICAL TRIAL: NCT00273390
Title: The Use of Remicade (Infliximab) in the Management of Vision-threatening Uveitis That is Refractory to Other Modes of Systemic Immunosuppression
Brief Title: A Clinical Trial of Infliximab for Uveitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Centocor, Inc. (Industry)
Other Study IDs: e1473
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2008-01

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis | interventions — Infliximab

INTERVENTIONS:
Drug: Remicade (infliximab)

SUMMARY:
This project is designed to test the hypothesis that inhibition of binding between tumor necrosis factor alpha (TNF-alpha) and its receptors using Remicade (infliximab, chimeric mouse/human IgG1K monoclonal antibody directed against human TNF-alpha, Centocor, Malvern,PA) is clinically useful for patients with uveitis that is refractory to other forms of systemic immunosuppressive therapy.

ELIGIBILITY:
Inclusion Criteria:

1. The study group will include patients suffering from treatment-resistant vision-threatening uveitis who attend the Uveitis Clinic at Casey Eye Institute.
2. We plan to enroll 32 patients.

Exclusion Criteria:

1. Patients with ocular or systemic infection.
2. Patients with the subtype of uveitis termed pars planitis who have MRI scan evidence of demyelination. There is a theoretical risk of adverse outcome of TNF-alpha inhibition on the clinical course of multiple sclerosis. Patients who suffer from pars planitis are at increased risk of developing multiple sclerosis.
3. Children under the age of 9.
4. Patients with known sensitivity to mouse proteins. Remicade is a chimeric protein with human and murine components.
5. Patients with history of cancer (exception- skin cancers which are curatively resected), organ transplantation (exception- cornea), recent drug or alcohol addiction, or inability to keep appointments.
6. Patients with other serious systemic diseases that could interfere with participation in the study.
7. It is specifically noted that pregnant women and nursing mothers will be excluded from this study.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32
Dates: Start 2001-08; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James T Rosenbaum, MD, Principal Investigator — Oregon Health and Science University; Eric B Suhler, MD, Study Director — Oregon Health and Science University; Justine Smith, MBBS, Phd, Study Director — Oregon Health and Science University

REFERENCES:
- [Result] Suhler EB, Smith JR, Wertheim MS, Lauer AK, Kurz DE, Pickard TD, Rosenbaum JT. A prospective trial of infliximab therapy for refractory uveitis: preliminary safety and efficacy outcomes. Arch Ophthalmol. 2005 Jul;123(7):903-12. doi: 10.1001/archopht.123.7.903. PMID 16009830
- [Derived] Suhler EB, Smith JR, Giles TR, Lauer AK, Wertheim MS, Kurz DE, Kurz PA, Lim L, Mackensen F, Pickard TD, Rosenbaum JT. Infliximab therapy for refractory uveitis: 2-year results of a prospective trial. Arch Ophthalmol. 2009 Jun;127(6):819-22. doi: 10.1001/archophthalmol.2009.141. No abstract available. PMID 19506209